CLINICAL TRIAL: NCT02868749
Title: Comparative Clinical, Histological and Ultrasound Pilot Study of Two Hyaluronic Acid Gel Fillers, Designed for Deep Injection, in Adipose Tissue
Brief Title: Histology and Ultrasound Pilot Study of HA Gels Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vandeputte, Joan, M.D. (Individual)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: BVL/JVL
Record Dates: First submitted 2016-07-27; First posted 2016-08-16 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Atrophy
Keywords: Hyaluronic Acid; histology; ultrasound; subcutaneous; adipose tissue
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic Acid filler 1 for deep injection (Experimental): Injection Session 1 of Hyaluronic Acid filler 1, 3 weeks to 4 months before the surgery
  Injection Session 2 of Hyaluronic Acid filler 1, 5 to 9 days before the surgery
  Interventions: Device: Hyaluronic Acid filler
- Hyaluronic Acid filler 2 for deep injection (Active Comparator): Injection Session 1 of Hyaluronic Acid filler 2, 3 weeks to 4 months before the surgery
  Injection Session 2 of Hyaluronic Acid filler 2, 5 to 9 days before the surgery
  Interventions: Device: Hyaluronic Acid filler

INTERVENTIONS:
Device: Hyaluronic Acid filler — Linear retrograde, subcutaneous injection of 0,5 ml of hyaluronic acid gel in one side of the abdomen or one breast, 3 weeks to 4 months before the surgery.
Device: Hyaluronic Acid filler — Linear retrograde, subcutaneous injection of 0,5 ml of hyaluronic acid gel in other side of the abdomen or other breast, 5 to 9 days before the surgery.

SUMMARY:
This study is a single-blind intra-individual comparative study to evaluate the short and medium term tissue response after the injection of 2 brands of hyaluronic acid gels (HA), designed for deep injection, that have been used for several years on a worldwide scale.

DETAILED DESCRIPTION:
The study will be disclosed to patients who present with an indication for either abdominoplasty or bilateral breast reduction with a Wise pattern skin excision (inverted T inframammary scar) Informed consent will be obtained from volunteers at their next consultation, during which the preoperative preparation is finalised and the surgery is booked.

Participants will receive injections for the first time three weeks to four months before the operation and for the second time five to nine days before the operation, in tissue that will be removed during the surgery.

In each session, through one single access point, a linear retrograde, subcutaneous injection will be performed with 0,5 ml of each of the studied hyaluronic acid gels, each in an opposite direction, each parallel to the skin surface.

Both sessions will be monitored by ultrasound examination. After the injections, the 2 cm of injected area which is most remote from the entrance point of the cannula will be remodelled by finger pressure and tissue pinching, to simulate remodelling as commonly performed after filler injection.

At the beginning of the operation, the injected subcutaneous fat will be removed with the overlying skin, to be sent for histologic examination.

The objective of the histologic examination is to assess the tissue response at one week versus three weeks to four months after the injection, as well as to assess the spread of the products, with and without remodelling after injection.

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for and requesting abdominoplasty
* patients eligible for and requesting bilateral breast reduction

Exclusion Criteria:

* Patients prone to hypertrophic scarring or keloids
* Hypersensitivity to hyaluronic acid
* Hypersensitivity to lidocaine or amide type local anaesthetics
* Autoimmune disease
* Severe, multiple allergies or anaphylactic shock
* Epilepsy
* Heart rhythm disorders
* Porphyria, congenital methemoglobinemia, glucose-6 phosphate dehydrogenase deficiencies, treatment with methaemoglobin-inducing substances.
* Previous streptococcal disease (acute rheumatic fever whether or not with heart valve involvement)
* Patients on medication which slows hepatic metabolism (such as cimetidine, beta-blockers)
* Diabetes requiring insulin treatment
* Major system disease.
* Coagulation disorders. Anticoagulation therapy. Chronic use of acetylsalicylic acid.
* Previous surgery in the areas eligible for injections.
* All contraindications to their surgical treatment (such as pregnancy or lactation).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
tissue inflammation after injection of hyaluronic acid filler | 3 weeks to 4 months after injection
  Presence of lymphocytes and/ or histiocytes around the filler through histologic examination [Yes/No]

SECONDARY OUTCOMES:
tissue response after injection of hyaluronic acid filler | 1 week after injection
  Presence of lymphocytes and/ or histiocytes and/ or macrophages around the filler through histologic examination [Yes/No]
tissue response after injection and remodelling of hyaluronic acid filler | 3 weeks to 4 months after injection
  Presence of lymphocytes and/ or histiocytes and/ or macrophages around the filler through histologic examination [Yes/No]
tissue response after injection and remodelling of hyaluronic acid filler | 1 week after injection
  Presence of lymphocytes and/ or histiocytes and/ or macrophages around the filler through histologic examination [Yes/No]
filler distribution in tissue | 3 weeks to 4 months after injection
  The height and width of the total filler spread [mm]
filler distribution in tissue | 1 week after injection
  The height and width of the total filler spread [mm]

CONTACTS AND LOCATIONS:
Overall Officials: Joan H Vandeputte, MD, Principal Investigator — A.Z Oudenaarde (Oudenaarde General Hospital)
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - A.Z. Oudenaarde, Oudenaarde

IPD SHARING:
Plan to Share IPD: Yes
pilot study on 5 patients: min, max, average measurements will be published

REFERENCES:
- [Background] Flynn TC, Sarazin D, Bezzola A, Terrani C, Micheels P. Comparative histology of intradermal implantation of mono and biphasic hyaluronic acid fillers. Dermatol Surg. 2011 May;37(5):637-43. doi: 10.1111/j.1524-4725.2010.01852.x. Epub 2011 Jan 27. PMID 21272119
- [Background] Hirsch RJ, Narurkar V, Carruthers J. Management of injected hyaluronic acid induced Tyndall effects. Lasers Surg Med. 2006 Mar;38(3):202-4. doi: 10.1002/lsm.20283. PMID 16485276
- [Background] Arlette JP, Trotter MJ. Anatomic location of hyaluronic acid filler material injected into nasolabial fold: a histologic study. Dermatol Surg. 2008 Jun;34 Suppl 1:S56-62; discussion S62-3. doi: 10.1111/j.1524-4725.2008.34244.x. PMID 18547183
- [Background] Micheels P, Sarazin D, Besse S, Sundaram H, Flynn TC. A blanching technique for intradermal injection of the hyaluronic acid Belotero. Plast Reconstr Surg. 2013 Oct;132(4 Suppl 2):59S-68S. doi: 10.1097/PRS.0b013e31829a02fb. PMID 24077012
- [Background] Franca Wanick FB, Almeida Issa MC, Luiz RR, Soares Filho PJ, Olej B. Skin Remodeling Using Hyaluronic Acid Filler Injections in Photo-Aged Faces. Dermatol Surg. 2016 Mar;42(3):352-9. doi: 10.1097/DSS.0000000000000659. PMID 26918965
- [Background] Shaw RB Jr, Katzel EB, Koltz PF, Kahn DM, Girotto JA, Langstein HN. Aging of the mandible and its aesthetic implications. Plast Reconstr Surg. 2010 Jan;125(1):332-342. doi: 10.1097/PRS.0b013e3181c2a685. PMID 20048624
- [Background] Rohrich RJ, Pessa JE. The fat compartments of the face: anatomy and clinical implications for cosmetic surgery. Plast Reconstr Surg. 2007 Jun;119(7):2219-2227. doi: 10.1097/01.prs.0000265403.66886.54. PMID 17519724
- [Background] Pilsl U, Rosmarin W, Anderhuber F. The premaxillary space: a location for filler injection? Dermatol Surg. 2014 Mar;40(3):301-4. doi: 10.1111/dsu.12431. Epub 2014 Jan 30. PMID 24479675